CLINICAL TRIAL: NCT00669695
Title: Systemic Inflammation and Obstructive Sleep Apnea Syndrome: Effect of Atorvastatin
Acronym: StatinflaSAS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Interim analysis performed without efficient results
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 0721; 2007-005286-35 (Registry Identifier: ID RCB)
Record Dates: First submitted 2008-04-21; First posted 2008-04-30 (Estimated); Last update posted 2013-09-24 (Estimated); Status verified 2013-09

CONDITIONS: Obstructive Sleep Apnea Syndrome
Keywords: statins; cardiovascular risk; Obstructive sleep apnea syndrome (OSAS) patients
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Hydroxymethylglutaryl-CoA Reductase Inhibitors

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Stat/CPAP (Placebo Comparator): Atorvastatin and CPAP treatments
  Interventions: Drug: Atorvastatin treatment; Other: CPAP device
- Stat/sham CPAP (Placebo Comparator): Atorvastatin and sham CPAP treatments
  Interventions: Drug: Atorvastatin treatment; Other: sham CPAP treatment
- Placebo/CPAP (Sham Comparator): Placebo and CPAP treatments
  Interventions: Other: CPAP device
- Placebo/sham CPAP (Active Comparator): Placebo and sham CPAP treatments
  Interventions: Other: sham CPAP treatment

INTERVENTIONS:
Drug: Atorvastatin treatment — Atorvastatin treatment: tablets of 40 mg Atorvastatin will be administered orally, respecting the dosage of 40 mg/day, for 6 months.
  Other Names: statin
  Arms: Stat/CPAP; Stat/sham CPAP
Other: CPAP device — This device consists in a nasal continuous positive airway pressure (CPAP). It will be applied 3 months after the beginning of drug treatment and for 3 months.
  Other Names: positive air way pressure
  Arms: Placebo/CPAP; Stat/CPAP
Other: sham CPAP treatment — This device consists in a sham CPAP. It will be applied 3 months after the beginning of drug treatment and for 3 months.
  Other Names: sham CPAP
  Arms: Placebo/sham CPAP; Stat/sham CPAP

SUMMARY:
The aim of this clinical trial is to evaluate the effect of Atorvastatin on the endothelial function improvement during the obstructive sleep apnea syndrome (OSAS) after 3 months of treatment, by a double-blind, randomized, placebo-controlled, multi-center study.

An interim analysis will be performed when 25 patients per group will be included.

DETAILED DESCRIPTION:
Secondary objectives of this clinical trial :

* To evaluate the effect of Atorvastatin in comparison with the placebo on the inflammation occurring during OSAS, after 3 months of treatment.
* To evaluate the effect of Atorvastatin in comparison with the placebo on the insulin-resistance associated to OSAS, after 3 months of treatment.
* To evaluate the effect of Atorvastatin in comparison with the placebo on the hypercholesterolemia associated to OSAS, after 3 months of treatment.
* To evaluate at 6 months, the effect of the continuous positive airway pressure (CPAP) + Atorvastatin association on the previously cited parameters, in comparison with Atorvastatin, CPAP and placebo.
* To measure the CPAP efficiency in comparison with sham CPAP in patients receiving the placebo, after 3 months of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Men or women > 18 years old
* Subjects diagnosed with OSAS (apnea/hypopnea index = AHI > 30/h)
* Subjects with clinical ATH from grade I or II controlled with mono-therapy(140<SAP<180 mmHg and 90<DAP<110 mmHg)

Exclusion Criteria:

* Patients with a history of prior stroke or coronary ischemic disease
* Chronic respiratory disease (PaO2 < 60 mmHg and/or PaCO2 > 45 mmHg)
* Lung disease
* Hypothyroidism
* Statin treatment
* Antihypertensive treatment with more than one drug
* Pregnant or lactating women
* Alcohol consumption > 3 units/day
* Treatment by itraconazole, ketoconazole, antiprotease, fibrates, antivitamin K, diltiazem, verapamil, erythromycin, clarithromycin, cyclosporin.
* Hypersensitivity to one of the drug compounds
* Patients with modified concomitant treatments during the 3 months before inclusion
* Potentially dangerous sleepiness
* Jobs at risk

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2008-05; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
The primary endpoint is the percent of peripheral arterial tone (PAT) improvement in comparison with the baseline situation. | after 3 months of Atorvastatin treatment.

SECONDARY OUTCOMES:
Evaluation of the inflammation occurring during OSAS. | after 3 months of Atorvastatin or placebo treatment.
Evaluation of the insulin-resistance associated to OSAS. | after 3 months of Atorvastatin or placebo treatment.
Evaluation of the hypercholesterolemia associated to OSAS. | after 3 months of Atorvastatin or placebo treatment.
Evaluation of the effect of continuous positive airway pressure (CPAP) + Atorvastatin association on the previously cited parameters, in comparison with effect of Atorvastatin, CPAP and placebo. | after 6 months of treatments
Measurement of the CPAP efficiency in comparison with sham CPAP in patients receiving the placebo. | after 3 months of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Louis PEPIN, MD, PhD, Principal Investigator — University Hospital of Grenoble, France
Locations (4):
- France (3):
  - Universitary Hospital of Angers, Angers
  - Hospital of Annemasse, Annemasse
  - University Hospital of Grenoble, Grenoble
- Universitary Hospital of Geneva, Geneva, Switzerland

REFERENCES:
- [Background] Bergeron C, Kimoff J, Hamid Q. Obstructive sleep apnea syndrome and inflammation. J Allergy Clin Immunol. 2005 Dec;116(6):1393-6. doi: 10.1016/j.jaci.2005.10.008. No abstract available. PMID 16337480
- [Derived] Jullian-Desayes I, Tamisier R, Zarski JP, Aron-Wisnewsky J, Launois-Rollinat SH, Trocme C, Levy P, Joyeux-Faure M, Pepin JL. Impact of effective versus sham continuous positive airway pressure on liver injury in obstructive sleep apnoea: Data from randomized trials. Respirology. 2016 Feb;21(2):378-85. doi: 10.1111/resp.12672. Epub 2015 Nov 16. PMID 26567858
- [Derived] Joyeux-Faure M, Tamisier R, Baguet JP, Dias-Domingos S, Perrig S, Leftheriotis G, Janssens JP, Trzepizur W, Launois SH, Stanke-Labesque F, Levy PA, Gagnadoux F, Pepin JL. Response to statin therapy in obstructive sleep apnea syndrome: a multicenter randomized controlled trial. Mediators Inflamm. 2014;2014:423120. doi: 10.1155/2014/423120. Epub 2014 Aug 25. PMID 25221387